CLINICAL TRIAL: NCT07110337
Title: A Prospective Study to Evaluate the Use of the Minder Device to Aid in Developing a Treatment Plan After Inconclusive Prolonged EEG in Patients With Epilepsy
Brief Title: Diagnosing Epilepsy To EffeCT Change
Acronym: DETECT
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Epiminder America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Diagnostic
Other Study IDs: EM2401
Record Dates: First submitted 2025-07-24; First posted 2025-08-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy; Epilepsy (Treatment Refractory)
Keywords: Minder System; Sub-scalp EEG monitoring device
MeSH Terms: conditions — Epilepsy | interventions — Electroencephalography; Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Minder System Treatment Arm (Experimental)
  Interventions: Device: Receipt of the Minder System (implantable sub-scalp continuous electroencephalographic (EEG) monitoring (iCEM) system)
- Minder System Control Arm (Placebo Comparator)
  Interventions: Device: Receipt of the Minder System (implantable sub-scalp continuous electroencephalographic (EEG) monitoring (iCEM) system)
- Standard of Care Arm (No Intervention)

INTERVENTIONS:
Device: Receipt of the Minder System (implantable sub-scalp continuous electroencephalographic (EEG) monitoring (iCEM) system) — The Minder System consists of an implanted device containing an electrode lead and telemetry unit. The electrode lead contains four electrodes that are placed under the patient's scalp to record electrical activity (EEGs) from both sides of the brain. The electrode lead is connected to the telemetry unit that continuously transmits these signals to the external Minder devices to remotely show EEGs for clinician review.
  Arms: Minder System Control Arm; Minder System Treatment Arm

SUMMARY:
The purpose of this research is to address the challenges of diagnosing and long-term management of epilepsy in participants whose seizures are not well captured by standard electroencephalography (EEG) tests and who cannot use or are not able to use more standard monitoring techniques. This research will compare the Minder System to standard of care in providing reliable seizure data. The Minder System was granted De Novo classification by the U.S. Food and Drug Administration (FDA) and is not investigational.

Participants will consent to join the study and be implanted with the Minder device; or consent to join the study and continue with their Standard of Care (SOC) as a control group. Participants chose to be implanted with the Minder device will have the device implanted under their scalp. After implantation, participants will be randomly assigned to a group where their treating physician will have access to the EEG data collected by the Minder System or a group where their treating physician does not have access to the EEG data collected by the Minder System. Participants receiving the Minder System will not know which group they are in (blinded) until the study ends.

All participants will continue to be followed by their treating physician and undergo assessments and visits until enough information is available to determine a treatment plan or the 6-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of focal and/or generalized epilepsy.
* Drug-resistant
* At least an average of 1 seizure within the past 3 months
* Participant completed a multi-day EEG assessment that was inconclusive, and is unchanged since the last EEG monitoring.

Exclusion Criteria:

* Epilepsy surgery within the past 6 months
* Active Deep Brain Stimulation (DBS) or Responsive Neurostimulator System (RNS)
* Participant needs treatments or assessments that are not indicated with the Minder System like Magnetic Resonance Imaging (MRI), Electro-Convulsive Therapy (ECT), lithrotripsy, and diathermy
* Participant cannot have surgery to have the device implanted

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Compare the proportion of participants receiving the Minder System with those receiving Standard of Care (SOC) as a means of obtaining an actionable event based on clinical data (i.e. Minder EEG data, non-Minder EEG data, SOC assessments, etc.). | 6 months

SECONDARY OUTCOMES:
Compare the time to the first actionable event. | 6 months
Compare participant wellbeing between groups with the Beck Depression Inventory (BDI) for symptoms associated with depression. | 6 months
Compare participant wellbeing between groups with the Beck Anxiety Inventory (BAI) for symptoms associated with anxiety. | 6 months
Compare healthcare utilization between groups by the number of hospital visits. | 6 months
Compare healthcare utilization between groups by medication usage. | 6 months
Compare healthcare utilization between groups by the number of surgeries or procedures. | 6 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - Mayo Clinic - Florida, Jacksonville, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Halliday AJ, Gillinder L, Lai A, Seneviratne U, Fontenot H, Cameron T, McLean K, Niemiec A, Raghupathi R, Ganguly TM, Ellis C, Conrad EC, Briggs R, Bulluss K, Kwan P, Perucca P, O'Brien TJ, McGonigal A, Gutman M, Papacostas J, Fong MWK, Lee A, Crompton DE, Laing J, Wijayath M, Morokoff AP, Murphy M, D'Souza WJ, Cook MJ. The UMPIRE study: A first-in-human multicenter trial of bilateral subscalp monitoring for epileptic seizure detection. Epilepsia. 2025 Sep;66(9):3426-3439. doi: 10.1111/epi.18458. Epub 2025 May 30. PMID 40445205